CLINICAL TRIAL: NCT00558948
Title: Musculoskeletal Outcomes After Bone Marrow Transplant
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Kathy Ruble, PhDc, RN, SKCCC
Other Study IDs: J06120; 1F31NR010038-01 (NIH)
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Survivors of Bone Marrow Transplant; Autologous and Allogeneic
Keywords: Bone Marrow Transplant; Bone Mineral Density; Survivors; Muscle Strength

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to evaluate bone mineral density and muscle strength in survivors of bone marrow transplant. Association with age, type of transplant, steroids, years since transplant, body composition, endocrinopathies, radiation, quality of life and physical activity will be explored.

DETAILED DESCRIPTION:
Bone marrow transplant survivors are at risk of diminished bone mineral density. Mechanisms and risks are not well understood. This study will help identify risks factors for developing this complication.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8-30 years
* One year from transplant

Exclusion Criteria:

* No current steroid use
* Medical conditions that would prohibit testing
* Neuropsychological conditions that prohibit completing questionnaires

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Survivors of bone marrow transplant (autologous and allogeneic) who are at least 1 year from transplant.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Ruble, PhDc, RN, Study Director — Johns Hopkins University, School of Nursing
Locations (1):
- Johns Hopkins University, Bayview Campus, Baltimore, Maryland, United States